CLINICAL TRIAL: NCT01308970
Title: Quantification of Outcome Measures for Mind-body Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, John W. Denninger, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2010P002785; R01AT006464 (NIH)
Record Dates: First submitted 2011-02-24; First posted 2011-03-04 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Stress, Psychological; Stress, Physiological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stress Management Group 1 (Experimental)
  Interventions: Behavioral: Stress Management Group 1
- Stress Management Group 2 (Experimental)
  Interventions: Behavioral: Stress Management Group 2
- Stress Management Group 3 (Experimental)
  Interventions: Behavioral: Stress Management Group 3

INTERVENTIONS:
Behavioral: Stress Management Group 1 — Subjects will attend individual stress management sessions once weekly for 8 weeks and will be instructed to listen to a health education CD for 20 minutes every day for the duration of the study.
  Arms: Stress Management Group 1
Behavioral: Stress Management Group 2 — Subjects will attend individual stress management sessions once weekly for 8 weeks and will be instructed to listen to a health education CD for 20 minutes every day for the duration of the study.
  Arms: Stress Management Group 2
Behavioral: Stress Management Group 3 — Subjects will attend individual stress management sessions once weekly for 8 weeks and will be instructed to listen to a health education CD for 20 minutes every day for the duration of the study.
  Arms: Stress Management Group 3

SUMMARY:
The purpose of this study is to determine if participation in one of three different health management groups will elicit genomic and biochemical changes and decrease perceived stress levels and symptoms in healthy, stressed adults. The investigators expect that changes in self-reported psychological stress and symptoms will be directly linked to changes in biological indicators (genomic expression profiles and neuroendocrine and pro-inflammatory biomarkers).

DETAILED DESCRIPTION:
This randomized, controlled trial will determine the relative strength of correlation between changes in stress outcome measures (self-report questionnaire, genomic expression, biochemical assay) in moderately to severely stressed healthy subjects randomized to one of three health education interventions at both end-intervention and at a 6-month long-term follow-up. This study will also determine which of the different outcome measures exhibit the greatest degree of sensitivity, reliability and consistency at both end-intervention and long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Stress is chronic and ongoing with no resolution of the stressors within the timeframe of the study, with a minimum prior duration of 6 months.
* Able to provide informed consent and to understand written and spoken English.

Exclusion Criteria:

* Practice of yoga, meditation, guided imagery or other mind body techniques that elicit the RR, once per week for 45 min total or more within the last three months or less.
* Any current medical condition that would preclude their safe and effective practice of the yoga or meditation interventions.
* The presence of bipolar or psychotic disorders, or history of any other DSMIV Axis I disorder with active symptoms or treatment within the last 5 years, as determined by a structured clinical interview.
* Initiation of psychotherapy within 6 months of entering the study.
* Serious or unstable medical illness, including serious or unstable cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease.
* Patient deemed unable to complete protocol due to cognitive, psychiatric or other reasons.
* Pregnancy or planned conception over the course of the study (could confound biomarker values).
* Current use of the following medications: systemic corticosteroids, chronic (i.e., more than 3 days per week) use of anti-inflammatories (e.g., ibuprofen; currently or within the last 3 months), immunosuppressive or cytotoxic therapies (currently or within the last 12 months), and anabolic steroids.
* Current (within the last 6 months) psychoactive medications (e.g. antidepressants, mood stabilizers, antipsychotics, anxiolytics), with the exception of hypnotics, which will be permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2011-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Levels Post-intervention and at 6-month Follow-up | Baseline (Week 1), Endpoint (Week 9), Follow-Up (Week 26)
  Perceived Stress Scale (PSS-10)
Change in Genomic Expression Profile Post-intervention and at 6-month Follow-up | Baseline (Week 1), Endpoint (Week 9), Follow-Up (Week 26)

CONTACTS AND LOCATIONS:
Overall Officials: John W Denninger, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Benson-Henry Institute for Mind Body Medicine; Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Denninger JW, Joss D, Romero PM, Khalsa SBS, Hoge EA, Bhasin M, Lazar SW, Dusek JA, Macklin E, Libermann T, Fricchione GL, Benson H. Psychological assessments, allostatic load and gene expression analyses in a randomized controlled trial comparing meditation, yoga, and stress education. Front Psychol. 2025 Sep 12;16:1653242. doi: 10.3389/fpsyg.2025.1653242. eCollection 2025. PMID 41020112